CLINICAL TRIAL: NCT06182098
Title: Value of Intravenous Fluids in the Emergent Treatment of Pediatric Migraine
Brief Title: Intravenous Fluids in Pediatric Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dayton Children's Hospital (Other)
Responsible Party: Principal Investigator, Jonathan Elliott, MD, Principal Investigator, Dayton Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-029
Record Dates: First submitted 2023-08-29; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Migraine; Migraine in Children
Keywords: migraine; headache; pediatric; fluids; bolus
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Saline Solution; Ketorolac; Ketorolac Tromethamine; Diphenhydramine; Prochlorperazine; NOP-bolus regimen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus (Experimental): Will receive a normal saline bolus
  Interventions: Drug: Ketorolac; Drug: Diphenhydramine; Drug: Prochlorperazine; Other: bolus
- Control (Placebo Comparator): Will receive 1/2 maintenance normal saline
  Interventions: Other: 1/2 maintenance fluids; Drug: Ketorolac; Drug: Diphenhydramine; Drug: Prochlorperazine

INTERVENTIONS:
Other: 1/2 maintenance fluids — Patients will receive 1/2 maintenance normal saline (with a maximum of 50 mL/hr), over one hour.
  Other Names: Normal saline
  Arms: Control
Drug: Ketorolac — 0.5mg/kg, with a maximum of 30mg
  Other Names: Toradol
Drug: Diphenhydramine — 0.5mg/kg, with a maximum of 25mg
  Other Names: Benadryl
Drug: Prochlorperazine — 0.15mg/kg, with a maximum of 10mg
  Other Names: Compazine
Other: bolus — 20mL/kg normal saline bolus, with a maximum of 1L, given over one hour
  Other Names: normal saline
  Arms: Bolus

SUMMARY:
The goal of this clinical trial is to compare intravenous (IV) fluids in pediatric patients with migraine. The main questions it aims to answer are:

* Does a large amount of fluids (bolus) improve pain
* Does a large amount of fluids (bolus) reduce admissions to the hospital for migraine Participants will be asked to report their pain and have vital signs checked every 30 minutes for two hours.

Researchers will compare a large amount of fluids (bolus) to a small amount (half maintenance) to see if there is a difference in pain improvement.

DETAILED DESCRIPTION:
Patients will be randomized to one of two treatment groups. The intervention group will receive a 20 mL/kg bolus of normal saline (with a maximum of 1L), given over one hour.

The control group will receive normal saline at half maintenance (with a maximum of 50mL/hr) over one hour.

Both groups will receive:

* ketoralac (Toradol), 0.5mg/kg, with a maximum of 30mg
* diphenhydramine(Benadryl), 0.5mg/kg, with a maximum of 25mg
* prochlorperazine(Compazine), 0.15mg/kg, with a maximum of 10mg

Pain score, heart rate, and blood pressure will be monitored every 30 minutes from the start of the medications/fluids being started, for a period of two hours. Pain will be recorded using a 100mm visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 prior headache
* Minimum pain score of 10mm
* Headache lasting 2-72 hours
* At least two of the following four: 1 Bifrontal/bitemporal or unilateral location, 2 Pulsating quality, 3 Moderate or severe pain intensity, 4 Aggravation by or causing avoidance of routine physical activity
* At least one of the following: 1 Nausea and/or vomiting, 2Photophobia and phonophobia, 3 Not better accounted for by another ICHD-3 diagnosis

Exclusion Criteria:

* Shunted hydrocephalus
* Temperature equal to or greater than 38.5C
* Clinical suspicion of meningitis
* Known or suspected intracranial lesion
* Clinical evidence of significant dehydration (or signs of shock, or attending discretion)
* Head trauma in previous 7 days
* Pregnancy or breastfeeding
* Initial pain score less than 10mm
* Allergy to study medications
* Patients previously participating in the study

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
One hour change in pain | one hour
  Mean change from baseline pain score, taken at one hour from beginning data collection. A 100 mm visual analog scale is used, with a higher score indicating higher pain. A greater change in pain score means more improved pain.

SECONDARY OUTCOMES:
Two hour change in pain | two hours
  Mean change from baseline pain score, taken at two hours from beginning of data collection. A 100 mm visual analog scale is used, with a higher score indicating higher pain. A greater change in pain score means more improved pain.
length of emergency stay | Through study completion, up to 24 hours after patient enrollment.
  Mean duration of emergency department visit, reported in hours.
return visits | Through study completion, up to 48 hours after completion of study protocol.
  percent of patients with additional visits to the emergency department within 48 hours of discharge
Admission rate | during emergency department visit, up to 24 hours after patient enrollment
  Percentage of patients admitted to the hospital for migraine
Resolution of pain | Through study completion, up to 24 hours after enrollment
  Percentage of patients with complete resolution of pain at the time of emergency discharge
50% reduction of pain | Through study completion, up to 24 hours after enrollment. Assessed at the time of discharge from the emergency department
  Percentage of patients with at least 50% reduction of pain from baseline, at the time of emergency discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Elliott, MD, Principal Investigator — Dayton Children's
Locations (1):
- Dayton Children's Hosptial, Dayton, Ohio, United States